CLINICAL TRIAL: NCT07333339
Title: Comparative Effects of BCI-Based Attention Training, Methylphenidate, and Citicoline on Attention and Executive Function in School-Age Children: A Naturalistic Quasi-Experimental Study
Brief Title: A Brain-Computer Interface-Based Attention Training Program Compared With Methylphenidate and Citicoline
Acronym: Brain-Computer
Status: Completed | Type: Observational
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Serkan Turan, Assoc Prof., Uludag University
Other Study IDs: THIZ-2023-1670
Record Dates: First submitted 2025-12-16; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD); Brain Computer Interface
Keywords: Brain-computer interface; attention training; methylphenidate; citicoline; cognitive training; executive functions
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 8 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- COGO + Methylphenidate: Children in this cohort receive a combined intervention consisting of a brain-computer interface (BCI)-based attention training program (COGO) together with methylphenidate prescribed as part of routine clinical care. The attention training is delivered through game-based computerized sessions that adapt to the child's attention-related brain signals. Methylphenidate dosing follows standard clinical practice and is determined by the treating clinician.
  Interventions: Device: Brain-Computer Interface-Based Attention Training
- COGO + Citicoline: Children in this cohort receive the same BCI-based attention training program (COGO) combined with citicoline supplementation. Citicoline is administered in age-appropriate doses as part of usual clinical care. The BCI training consists of structured, game-based sessions designed to support sustained attention and cognitive control.
  Interventions: Device: Brain-Computer Interface-Based Attention Training
- COGO Only: Children in this cohort participate only in the BCI-based attention training program (COGO), without concurrent stimulant medication or citicoline supplementation. The training is delivered through computerized, game-based sessions that adjust task demands based on real-time attention-related brain signals.
  Interventions: Device: Brain-Computer Interface-Based Attention Training
- Citicoline Only: Children in this cohort receive citicoline supplementation alone, without participation in the BCI-based attention training program. Citicoline is administered in age-appropriate doses as part of routine clinical management for attention-related difficulties.
  Interventions: Device: Brain-Computer Interface-Based Attention Training

INTERVENTIONS:
Device: Brain-Computer Interface-Based Attention Training — The intervention consists of a brain-computer interface (BCI)-based attention training program delivered through computerized, game-based tasks that adapt in real time to the participant's attention-related brain activity recorded via EEG. Task difficulty and progression are dynamically adjusted based on neural markers of attentional engagement, creating a closed-loop training environment designed to support sustained attention, response control, and executive functioning.
  In some participants, this training is used in combination with pharmacological or nutraceutical support as part of routine clinical care. Methylphenidate is prescribed according to standard pediatric clinical guidelines and individualized clinical judgment. Citicoline is administered in age-appropriate doses as a nutritional supplement intended to support cognitive and neural functioning. No experimental dosing or protocol-driven medication adjustments are applied.
  All interventions are delivered in a naturalistic

SUMMARY:
The goal of this observational study is to learn whether a brain-computer interface (BCI)-based attention training program, used alone or together with medication, can improve attention, executive functioning, and emotional regulation in school-age children with attention difficulties.

The study focuses on school-age children who were referred for problems with attention, concentration, or related cognitive and emotional difficulties.

The main questions it aims to answer are:

Does BCI-based attention training improve children's attention and response control when used on its own?

Do children show greater improvements when BCI-based attention training is combined with medication such as methylphenidate or citicoline?

Are there differences in attention, executive functioning, or emotional symptoms between children receiving combined approaches versus single treatments?

Researchers compared four naturally occurring treatment approaches to see whether combining attention training with medication leads to better outcomes than using one method alone.

Participants will:

Take part in a computerized, game-based BCI attention training program that uses brain signals to guide training tasks

Receive medication (methylphenidate or citicoline) if this was part of their usual clinical care

Complete computerized attention tests that measure focus, reaction time, and impulse control

Have parents complete questionnaires about attention, behavior, emotions, and everyday executive functioning before and after the intervention

This study was conducted in a real-world clinical setting and reflects routine treatment choices made by families and clinicians, rather than random assignment. The findings aim to help families and health care providers better understand how different treatment combinations may support attention and self-regulation in children.

DETAILED DESCRIPTION:
Attention difficulties in childhood, including problems with sustained focus, impulse control, and executive functioning, are common reasons for referral to child and adolescent mental health services. While stimulant medications such as methylphenidate are widely used and effective for many children, not all families prefer medication alone, and some children continue to experience cognitive or emotional difficulties despite treatment. For these reasons, there is growing interest in non-pharmacological and combined approaches that target attention through different mechanisms.

One emerging approach is brain-computer interface (BCI)-based attention training. These programs use real-time brain signals, recorded through EEG sensors, to adapt game-like tasks that encourage sustained attention and cognitive control. Unlike traditional computer games, task difficulty and progression change dynamically based on the child's level of attentional engagement. This makes training more interactive and potentially more closely linked to underlying brain processes involved in attention regulation.

In routine clinical practice, some children receive BCI-based attention training alone, while others use it together with medication such as methylphenidate or citicoline. Citicoline is a nutritional supplement that has been suggested to support brain function and cognitive processes, although evidence in children remains limited. How these different approaches compare with one another, and whether combining them offers added benefit, is still not well understood.

This study was conducted in a naturalistic clinical setting, meaning that treatment choices were made as part of usual care rather than through random assignment. Children were grouped based on the intervention they received: BCI-based attention training alone, BCI combined with methylphenidate, BCI combined with citicoline, or citicoline alone. All children completed standardized assessments before and after the intervention period.

Attention and cognitive performance were evaluated using a computerized continuous performance test that measures sustained attention, reaction time, variability of responses, and impulse control. In addition, parents completed validated questionnaires assessing attention-related symptoms, emotional difficulties, and everyday executive functioning such as planning, inhibition, and emotional regulation.

By examining changes within each treatment group and comparing overall patterns across groups, this study aims to provide clinically meaningful information about how different treatment strategies may support attention and self-regulation in children. The findings are intended to help families and health care providers make more informed decisions about combining digital attention training with medication in real-world clinical settings.

ELIGIBILITY:
Inclusion Criteria:

School-age children (approximately 6-18 years)

Clinical diagnosis of Attention-Deficit/Hyperactivity Disorder (ADHD)

Presence of attention or executive-function difficulties requiring clinical follow-up

Participation in one of the routine clinical interventions (BCI-based attention training, methylphenidate, citicoline, or their combination)

Completion of baseline and post-intervention assessments

Written informed consent obtained from a parent or legal guardian

Exclusion Criteria:

Presence of a neurological disorder (e.g., epilepsy, traumatic brain injury)

Intellectual disability or severe developmental disorder that would prevent participation in computerized assessments

Current use of additional psychotropic medications other than methylphenidate

Significant sensory or motor impairment interfering with computer-based testing

Incomplete assessment data or inability to complete the intervention period

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population consists of school-age children referred to a child and adolescent psychiatry outpatient clinic due to attention-related difficulties. All participants have a clinical diagnosis of Attention-Deficit/Hyperactivity Disorder (ADHD) and were receiving routine clinical care at the time of enrollment. The population reflects a real-world clinical sample, including children with varying levels of attentional, executive-function, and emotional difficulties commonly observed in pediatric ADHD. Treatment selection was based on usual clinical decision-making rather than random assignment.
Sampling Method: Non-Probability Sample
Enrollment: 174 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2025-11-10 (Actual)

PRIMARY OUTCOMES:
Conners Continuous Performance Test-Third Edition (CPT-3) | 8 weeks
  Outcome Measure 1:Conners Continuous Performance Test-Third Edition CPT-3)-Omission Errors.Number of omission errors reflecting inattention, reported as standardized T-scores based on CPT-3 normative data.Unit of Measure: T-score.
  Outcome Measure 2:CPT-3-Commission Errors. Number of commission errors reflecting impulsivity (standardized T-scores derived from CPT-3 normative data).Unit of Measure: T-score.
  Outcome Measure 3:CPT-3-Perseverations.Number of perseverative responses reflecting response control difficulties, reported as standardized T-scores based on CPT-3 normative data.Unit of Measure: T-score.
  Outcome Measure 4:CPT-3-Hit Reaction Time(HRT).Mean reaction time for correct responses (standardized T-scores derived from CPT-3 normative data).Unit of Measure: T-score.
  Outcome Measure 5:CPT-3-Hit Reaction Time Standard Deviation(HRT SD).Variability of reaction time across correct responses, reported as standardized T-scores based on CPT-3 normative data.Unit of Measure: T-score.

SECONDARY OUTCOMES:
1. Swanson, Nolan, and Pelham Rating Scale-Fourth Edition (SNAP-IV) | 8 weeks
  Description:
  The Swanson, Nolan, and Pelham Rating Scale-Fourth Edition (SNAP-IV) is a parent- or teacher-rated scale assessing symptoms of inattention, hyperactivity/impulsivity, and oppositional defiant behavior. Items are rated on a 4-point Likert scale (0-3), with higher scores indicating greater symptom severity.
  Score Range:
  Item scores range from 0 to 3; subscale scores are calculated as mean scores ranging from 0 to 3.
  Direction of Outcome:
  Higher scores indicate worse outcomes (greater symptom severity).
  Outcome Measure: Change in SNAP-IV total score from baseline to post-intervention.
2. Barkley Sluggish Cognitive Tempo Scale | 8 weeks
  Description:
  The Barkley Sluggish Cognitive Tempo Scale is a parent- or teacher-rated questionnaire assessing sluggish cognitive tempo symptoms, including excessive daydreaming, mental confusion, lethargy, and slowed behavior.
  Minimum-Maximum Score Range:
  Items are rated on a 4-point Likert scale ranging from 0 (never or rarely) to 3 (very often). Total and mean scores range from 0 to 3.
  Direction of Outcome:
  Higher scores indicate greater symptom severity and therefore worse outcomes.
  Outcome Measure: Change in Barkley SCT total score from baseline to post-intervention.
3. Revised Child Anxiety and Depression Scale (RCADS), Parent Version | 8 weeks
  Description:
  The Revised Child Anxiety and Depression Scale (RCADS) - Parent Form is a parent-rated questionnaire consisting of 47 items, assessing symptoms of anxiety and depression in children and adolescents across multiple DSM-based subscales (separation anxiety, social phobia, generalized anxiety, panic disorder, obsessive-compulsive disorder, and major depressive disorder).
  Minimum-Maximum Score Range:
  Items are rated on a 4-point Likert scale ranging from 0 (never) to 3 (always). Subscale and total raw scores range from 0 to 141. Raw scores may be converted to age- and sex-adjusted T-scores.
  Direction of Outcome:
  Higher scores indicate greater anxiety and depressive symptom severity and therefore worse outcomes.
  Outcome Measure: Change in RCADS total score from baseline to post-intervention.
4. Strengths and Difficulties Questionnaire (SDQ) | 8 weeks
  Description:
  The Strengths and Difficulties Questionnaire (SDQ) is a parent-rated behavioral screening questionnaire consisting of 25 items, assessing emotional symptoms, conduct problems, hyperactivity/inattention, peer relationship problems, and prosocial behavior in children and adolescents.
  Minimum-Maximum Score Range:
  Items are rated on a 3-point Likert scale ranging from 0 (not true) to 2 (certainly true). The Total Difficulties Score (sum of four difficulty subscales) ranges from 0 to 40. The Prosocial Behavior subscale ranges from 0 to 10.
  Direction of Outcome:
  For the Total Difficulties Score, higher scores indicate greater behavioral and emotional difficulties (worse outcomes). For the Prosocial Behavior subscale, higher scores indicate better outcomes.
  Outcome Measure: Change in SDQ Total Difficulties score from baseline to post-intervention.
5. Behavior Rating Inventory of Executive Function (BRIEF) | 8 weeks
  Description:
  The Behavior Rating Inventory of Executive Function (BRIEF) is a parent-rated questionnaire consisting of 86 items, designed to assess executive functioning in everyday settings in children and adolescents. It yields index scores including the Behavioral Regulation Index (BRI), Metacognition Index (MI), and a Global Executive Composite (GEC).
  Minimum-Maximum Score Range:
  Items are rated on a 3-point Likert scale. Raw scores are converted to age- and sex-adjusted T-scores, which typically range from 30 to 100.
  Direction of Outcome:
  Higher T-scores indicate greater executive function difficulties and therefore worse outcomes.
  Outcome Measure: Change in BRIEF Global Executive Composite T-score from baseline to post-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Serkan Turan, Principal Investigator — Uludag University
Locations (1):
- Uludag University, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared, as the data were collected in a naturalistic clinical setting and include sensitive health information. De-identified aggregate data may be reported in publications.

REFERENCES:
- [Background] 1. da Silva, B. S., Grevet, E. H., Silva, L. C. F., Ramos, J. K. N., Rovaris, D. L., & Bau, C. H. D. (2023). An overview on neurobiology and therapeutics of attention-deficit/hyperactivity disorder. Discover mental health, 3(1), 2. https://doi.org/10.1007/s44192-022-00030-1 2. Hwang, S., Meffert, H., Parsley, I., Tyler, P. M., Erway, A. K., Botkin, M. L., Pope, K., & Blair, R. J. R. (2019). Segregating sustained attention from response inhibition in ADHD: An fMRI study. NeuroImage. Clinical, 21, 101677. https://doi.org/10.1016/j.nicl.2019.101677 3. Noah, A.A., Sedky, H.E. New frontiers in pharmacological treatment of attention-deficit hyperactivity disorder. Naunyn-Schmiedeberg's Arch Pharmacol 398, 15025-15035 (2025). https://doi.org/10.1007/s00210-025-04328-z 4. Levy, F., Pipingas, A., Harris, E. V., Farrow, M., & Silberstein, R. B. (2018). Continuous performance task in ADHD: Is reaction time variability a key measure?. Neuropsychiatric disease and treatment, 14, 781-786. https://doi.org/10.2147/NDT.S158308 5. Kansakar, U., Trimarco, V., Mone, P., Varzideh, F., Lombardi, A., & Santulli, G. (2023). Choline supplements: An update. Frontiers in endocrinology, 14, 1148166. https://doi.org/10.3389/fendo.2023.1148166 6. Hübner, I. B., Scheibe, D. B., Marchezan, J., & Bücker, J. (2024). Use of Citicoline in Attention-Deficit/Hyperactivity Disorder: A Pilot Study. Clinical neuropharmacology, 47(5), 146-149. https://doi.org/10.1097/WNF.0000000000000602 7. Ölçüoğlu R. (2025). Neurofeedback for ADHD: Exploring the Role of Quantitative EEG and Brainwave Modulation. Brain and behavior, 15(8), e70714. https://doi.org/10.1002/brb3.70714 8. Jeunet, C., Glize, B., McGonigal, A., Batail, J. M., & Micoulaud-Franchi, J. A. (2019). Using EEG-based brain computer interface and neurofeedback targeting sensorimotor rhythms to improve motor skills: Theoretical background, applications and prospects. Neurophysiologie clinique = Clinical neurophysiology, 49(2), 125-136. https://doi.org/10.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-12-16): https://cdn.clinicaltrials.gov/large-docs/39/NCT07333339/Prot_SAP_000.pdf
  • Informed Consent Form (2025-12-16): https://cdn.clinicaltrials.gov/large-docs/39/NCT07333339/ICF_001.pdf